CLINICAL TRIAL: NCT00540436
Title: Study AMB107816, Clinical Evaluation of GSK1325760A in the Treatment of Pulmonary Arterial Hypertension (PAH)- An Open-Label Phase II/III Study to Evaluate the Efficacy, Safety and Pharmacokinetics of GSK1325760A -<Classification: Exploratory and Confirmatory Clinical Trial>
Brief Title: Evaluate the Efficacy, Safety and Pharmacokinetics of GSK1325760A in the Treatment of Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB107816
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2009-11-10 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Hypertension, Pulmonary
Keywords: Ambrisentan; Pulmonary Arterial Hypertension; 6MWD
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — ambrisentan

ARMS (1):
- GSK1325760A (Experimental): Single arm safety and efficacy
  Interventions: Drug: GSK1325760A

INTERVENTIONS:
Drug: GSK1325760A — Primary evaluation period: 5 mg/day, po, 12 weeks. Dose adjustment period: 2.5 mg, 5 mg or 10 mg/day, po, 12 weeks.
  Other Names: Ambrisentan

SUMMARY:
The primary objective of this study is to evaluate the effect of GSK1325760A on improvement in exercise capacity in subjects with pulmonary arterial hypertension (PAH).

The secondary objectives of this study are to evaluate administration of GSK1325760A on:

* The safety and tolerability
* Improvement of PAH
* The steady-state plasma pharmacokinetics of GSK1325760A

ELIGIBILITY:
Inclusion criteria:

* Subjects must have a diagnosis of Pulmonary Arterial Hypertension (PAH) in clinical classification of Pulmonary Hypertension Group1
* The mean right heart catheterization parameters measured from 6 months prior to the administration of the investigational drug must meet the criteria below:
* Mean pulmonary arterial pressure (mPAP) of >25 mmHg
* Pulmonary vascular resistance (PVR) of >3 mmHg/L/min
* Mean pulmonary capillary wedge pressure or left ventricular end diastolic pressure of <15 mmHg (if measurable)
* The measured six minutes walk distance (6MWD) at screening visit is in the range of =>150m and <=450m

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Japan (11):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Background] Yoshida S, Shirato K, Shimamura R, Nakahara N, Iwase T, Nakajima H. Efficacy, safety, and pharmacokinetics of ambrisentan in Japanese adults with pulmonary arterial hypertension. Curr Med Res Opin. 2011 Sep;27(9):1827-34. doi: 10.1185/03007995.2011.605440. Epub 2011 Aug 4. PMID 21812736

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK1325760A: First Treatment Period: GSK1325760A 5 mg once a day. Second Treatment Period: GSK1325760A 10 mg once a day (the dosage could be increased or decreased appropriately according to a participant's condition).
Period: First 12-Week Treatment Period
Arm/Group | GSK1325760A
Started | 25
Completed | 22
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Initiation of prohibited medication | 1
Period: Second 12-Week Treatment Period
Arm/Group | GSK1325760A
Started | 22
Completed | 21
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1325760A: GSK1325760A 5 mg once a day by Week 12. After Week 12, GSK1325760A 10 mg once a day (the dosage could be increased or decreased appropriately according to a participant's condition).
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (13.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese Heritage | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Six Minutes Walk Distance (6MWD) at Week 12
Description: Mean change from baseline was calculated as the Week 12 value minus the baseline value. 6MWD was measured by a 6 minute walk test. This test measures the distance that a subject can walk in a period of 6 minutes.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS): all participants registered, with the exception of those who had not received any dose of the investigational product and those who had no efficacy assessment after administration of the investigational product. Imputation technique was last observation carried forward.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
Meters | 33.49 (43.236)
Statistical Analysis 1: Comparison: GSK1325760A; Test type: Superiority or Other; Mean change = 33.49, 95% CI [15.231 to 51.744]

2. Secondary Outcome: Mean Change From Baseline in Six Minutes Walk Distance (6MWD) at Week 24/Withdrawal
Description: Change from baseline was calculated as the Week 24/Withdrawal value minus the basline value. 6MWD was measured by a 6 minute walk test. This test measures the distance that a subject can walk in a period of 6 minutes. Imputation technique was last observation carried forward.
Time Frame: Baseline and Week 24/Withdrawal
Population: Full Analysis Set
Measure: Median (Standard Deviation); unit: Meters
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
Meters | 46.82 (52.705)
Statistical Analysis 1: Comparison: GSK1325760A; Test type: Superiority or Other; Mean change = 46.82, 95% CI [24.566 to 69.076]

3. Secondary Outcome: Mean Change From Baseline in the Borg Dyspnea Index (BDI) at Weeks 12 and 24
Description: The BDI was calculated by using a 10-point scale (0 = None, 10 = Maximum). Change from baseline was calculated as the Week 12 and 24 values minus the baseline values. The BDI indicates the degree of breathlessness after completion of the 6 minute walk test. The BDI scale was assessed by each participant. Imputation technique was last observation carried forward.
Time Frame: Baseline and Weeks 12 and 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
Points on a scale
  Week 12 | -0.60 (2.157)
  Week 24 | -0.69 (1.904)

4. Secondary Outcome: Number of Participants With a Change From Baseline in Their World Health Organization (WHO) Functional Classification (FC) at Weeks 12 and 24
Description: There are four grades for WHO FC (class I = none, Class IV = most severe). The WHO FC indicates the severity of Pulmonary Arterial Hypertension and is an adaptation of the New York Heart Association classification. It was assessed by the investigator. Imputation technique was last observation carried forward.
Time Frame: Weeks 12 and 24
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
Participants
  Improved at Week 12 | 9
  No change at Week 12 | 16
  Deteriorated at Week 12 | 0
  Improved at Week 24 | 10
  No change at Week 24 | 14
  Deteriorated at Week 24 | 1

5. Secondary Outcome: Number of Participants With the Indicated Event, as an Assessment of Time to Clinical Worsening of Pulmonary Arterial Hypertension (PAH) at Week 24, Assessed as the First Occurrence of a Particular Event
Description: Time to clinical worsening is defined as the time from baseline to the first occurrence of death, lung transplantation, hospitalization for PAH treatment, atrial septostomy, or study discontinuation due to change to other PAH treatment. Time to clinical worsening is measured as the number of participants who experienced these events during 24 weeks.
Time Frame: Week 24
Population: Full Analysis Set: : all participants registered, with the exception of those who had not received any dose of the investigational product and those who had no efficacy assessment after administration of the investigational product
Measure: Number; unit: Participants
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
Participants
  Death | 0
  Lung transplantation | 0
  Hospitalization for PAH treatment | 0
  Atrial Septostomy | 0
  Study discontinuation (additional medication) | 1

6. Secondary Outcome: Mean Change From Baseline in Mean Pulmonary Atery Pressure (mPAP) and Mean Right Atrial Pressure (mRAP) at Weeks 12 and 24
Description: mPAP and mRAP are measures of cardiopulmonary hemodynamics. Change from baseline was calculated as the Week 12 and 24 values minus the baseline value. Observed data analysis (no imputation techniques).
Time Frame: Baseline and Weeks 12 and 24
Population: Full Analysis Set: Analysis was conducted using observed data only. Some participants were withdrawn before Week 24, or some participants could not be measured at Week 24 in this study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
mmHg
  mPAP (mmHg) at Week 12, n=21 | -6.29 (11.201)
  mRAP (mmHg) at Week 12, n=21 | -1.12 (3.761)
  mPAP (mmHg) at Week 24, n=16 | -8.69 (13.903)
  mRAP (mmHg) at Week 24, n=16 | -0.69 (3.683)

7. Secondary Outcome: Mean Change From Baseline in Cardiac Index (CI) at Weeks 12 and 24
Description: CI is a measure of cardiopulmonary hemodynamics. Change from baseline was calculated as the Week 12 and 24 values minus the baseline value. Observed data analysis (no imputation techniques).
Time Frame: Baseline and Weeks 12 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
L/min/m2
  Week 12, n=21 | 0.623 (0.5980)
  Week 24, n=16 | 0.598 (0.6115)

8. Secondary Outcome: Mean Change From Baseline in Cardiac Output (CO) at Weeks 12 and 24
Description: CO is a measure of cardiopulmonary hemodynamics. Change from baseline was calculated as the Week 12 and 24 values minus the baseline value. Observed data analysis (no imputation techniques).
Time Frame: Baseline and Weeks 12 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
L/min
  Week 12, n=21 | 1.033 (0.8783)
  Week 24, n=16 | 1.035 (0.9968)

9. Secondary Outcome: Mean Change From Baseline in Pulmonary Vascular Resistance (PVR) at Weeks 12 and 24
Description: PVR is a measure of cardiopulmonary hemodynamics. Change from baseline was calculated as the Week 12 and 24 values minus the baseline value. Observed data analysis (no imputation techniques).
Time Frame: Baseline and Weeks 12 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg/L/min
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
mmHg/L/min
  Week 12, n=21 | -7.257 (7.4344)
  Week 24, n=16 | -8.349 (7.6391)

10. Secondary Outcome: Mean Change From Baseline in B-type Natriuretic Peptide (BNP) Values at Weeks 12 and 24
Description: Change from baseline was calculated as the Week 12 and 24 values minus the baseline value. BNP is a surrogate maker of heart failure and was measured by a central laboratory. Observed data analysis (no imputation techniques).
Time Frame: Baseline and Weeks 12 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Nanograms/Liter (ng/L)
Arm/Group | GSK1325760A
Number analyzed (Participants) | 25
Nanograms/Liter (ng/L)
  Week 12, n=21 | -76.86 (160.942)
  Week 24, n=24 | -60.15 (248.345)

ADVERSE EVENTS:
Arm/Group | GSK1325760A
Serious Adverse Events (participants affected / at risk) | 4
Other Adverse Events (participants affected / at risk) | 24
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | GSK1325760A
Right ventricular failure (Cardiac disorders) | 2/25
Bacterial infection (Infections and infestations) | 1/25
Pneumonia (Infections and infestations) | 1/25
Pyelonephritis (Infections and infestations) | 1/25
Leukopenia (Blood and lymphatic system disorders) | 1/25
Vitreous hemorrhage (Eye disorders) | 1/25
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/25
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/25
Rash (Skin and subcutaneous tissue disorders) | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | GSK1325760A
Headache (Nervous system disorders) | 10/25
Nasopharyngitis (Infections and infestations) | 7/25
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5/25
Hot flush (Vascular disorders) | 4/25
Edema peripheral (General disorders) | 4/25
Anemia (Blood and lymphatic system disorders) | 3/25
Dizziness (Nervous system disorders) | 3/25
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3/25
Flushing (Vascular disorders) | 3/25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/25
Rash (Skin and subcutaneous tissue disorders) | 3/25
Blood pressure decreased (Investigations) | 2/25
Cystitis (Infections and infestations) | 2/25
Fatigue (General disorders) | 2/25
Insomnia (Psychiatric disorders) | 2/25
Leukopenia (Blood and lymphatic system disorders) | 2/25
Palpitations (Cardiac disorders) | 2/25
Somnolence (Nervous system disorders) | 2/25
Constipation (Gastrointestinal disorders) | 2/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.